CLINICAL TRIAL: NCT00280020
Title: Aging: Cytokine Mechanisms and Treatment of Insomnia
Brief Title: Behavioral Treatment of Insomnia in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Irwin, M.D., Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0061; R01AG026364 (NIH)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Aging; Insomnia
Keywords: sleep disorders; meditation; cognitive behavior therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavior Therapy (CBT)
- TCC (Experimental)
  Interventions: Behavioral: Tai Chi Chih (TCC)
- SS (Active Comparator)
  Interventions: Behavioral: Sleep Seminar (SS)

INTERVENTIONS:
Behavioral: Tai Chi Chih (TCC) — Participants will learn and practice 20 movements in 1 hour sessions twice per week for 16 weeks
  Arms: TCC
Behavioral: Cognitive Behavior Therapy (CBT) — For each 2-hour session held once a week for 16 weeks, the CBT treatment manual will outline objectives, patient skills, and treatment activities. Therapists will direct role-playing and other skill-development exercises that will be designed to increase patients' self-efficacy in managing their insomnia. Homework assignments will be planned weekly to ensure practice and skill application.
  Arms: CBT
Behavioral: Sleep Seminar (SS) — Each 2-hour session, held once a week for 16 weeks, consists of a 60-minute video presentation followed by a 60-minute question-and-answer discussion.
  Arms: SS

SUMMARY:
The purpose of this study is to evaluate whether Tai Chi Chih vs. cognitive behavioral therapy vs. sleep education reduces insomnia in older adults. The secondary goal of the study is to determine whether the behavioral treatment of insomnia alters proinflammatory cytokine activity.

DETAILED DESCRIPTION:
Insomnia is a prominent complaint in late-life. However, little scientific effort has been directed toward identifying the biological mechanisms that are related to abnormal sleep or to evaluating the efficacy of behavioral treatments for insomnia in older adults. Basic observations demonstrate that proinflammatory cytokines play a key role in the regulation of sleep. Previous research shows that cytokines are reciprocally linked with abnormal sleep. This trial builds upon these findings and extends a program of study that has examined the efficacy of behavioral interventions on health outcomes in the elderly.

Preliminary studies found that Tai Chi Chih (TCC), a slow moving meditation, contributes to improvements in subjective sleep quality, sleep amounts and sleep efficiency, alterations in sympathetic activity, decreases in proinflammatory cytokines, and improvements in health functioning in community-dwelling older adults. Additionally, cognitive behavior therapy (CBT) confers benefits on sleep outcomes.

In this randomized, controlled trial, 150 older adults will be randomly assigned to CBT, TCC, or sleep hygiene/education control (EC) over 16 weeks and followed for one year. The aims of this project are to: 1) evaluate the effects of CBT vs TCC vs. EC on objective and subjective measures of sleep and on fatigue, mood, and health functioning in older adults with insomnia; 2) determine the effects of CBT vs.TCC vs. EC on measures of proinflammatory cytokine activity and sympathovagal balance, and whether these two biological mechanisms are related to changes of disordered sleep over the course of the treatment trial; and 3) evaluate whether circulating levels of proinflammatory cytokines are associated with measures of sleep continuity in older adults with insomnia over the treatment trial. This study will advance psychobiological models of disordered sleep and the potential benefits of two readily exportable behavioral interventions for promoting improvements in sleep outcomes in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Older than 55 years of age at time of entry
* Sleep-onset delay, maintenance insomnia, or terminal insomnia
* Difficulties with sleep for a minimum of 3 nights per week
* Insomnia duration of at least 6 months
* Complaint of at least 1 negative effect during waking hours (e.g., fatigue, impaired functioning, mood disturbances) attributed to insomnia
* Habitual sleep-wake schedule reporting "lights-out" between 9:00 PM and midnight
* Accessible geographically

Exclusion Criteria:

* Evidence that insomnia is directly related to a medical disorder (e.g., hyperthyroidism) or effects of a medication that affects sleep structure and/or immune functioning
* Presence of sleep apnea or periodic limb movements during sleep
* Presence of another sleep disorder (e.g., Advanced or Delay Sleep Phase Syndrome)
* Regular use of a hypnotic or psychotropic medication (sleeping pills) and/or current psychotherapy or other behavioral therapy that would confound CBT or TCC
* Current history of a major psychiatric disorder (e.g. current major depression, alcohol or substance dependence, anxiety disorder)
* Cognitive impairment as suggested by a score lower than 23 on the Mini-Mental State examination
* Abnormal screening laboratory tests (e.g., abnormal thyroid hormone, elevated TSH, positive screening for HIV or hepatitis C)
* Smokers will also be excluded because of potential confounding effects on markers of inflammation
* Body mass index that is greater than 30 kg/m2 as obesity is associated with excessive levels of inflammatory markers
* Women must be post-menopausal
* Unable to commit to intervention schedule

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in insomnia symptoms as measured by subjective report and objective polysomnography | Subjective report: Baseline, 8, 12, 16 weeks, 3 months 1 year; PSG: Baseline, 16 weeks

SECONDARY OUTCOMES:
Changes in measures of proinflammatory cytokine activity. | Baseline, 8, 12, 16 weeks, 3 months 1 year (single samples); repeated blood sampling during PSG nights for circadian cytokine activity: Baseline, 16 weeks
Change in daytime impairment secondary to insomnia | Baseline, 8, 12, 16 weeks, 3 months 1 year
Changes in fatigue, depression and mood, and health function | Baseline, 8, 12, 16 weeks, 3 months 1 year
Changes in sympathovagal function and energy balance | Baseline, 8, 12, 16 weeks, 3 months 1 year
Changes in measures of interpersonal resilience and social | Baseline, 8, 12, 16 weeks, 3 months 1 year
Allostatic load | baseline, post-treatment, and one year follow-up
  CBC, glucose, HbA1c, lipids, fibrinogen, measures of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Irwin, MD, Principal Investigator — Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Irwin M, Pike J, Oxman M. Shingles Immunity and Health Functioning in the Elderly: Tai Chi Chih as a Behavioral Treatment. Evid Based Complement Alternat Med. 2004 Dec;1(3):223-232. doi: 10.1093/ecam/neh048. Epub 2004 Dec 1. PMID 15841255
- [Background] Irwin MR, Pike JL, Cole JC, Oxman MN. Effects of a behavioral intervention, Tai Chi Chih, on varicella-zoster virus specific immunity and health functioning in older adults. Psychosom Med. 2003 Sep-Oct;65(5):824-30. doi: 10.1097/01.psy.0000088591.86103.8f. PMID 14508027
- [Background] Motivala SJ, Sarfatti A, Olmos L, Irwin MR. Inflammatory markers and sleep disturbance in major depression. Psychosom Med. 2005 Mar-Apr;67(2):187-94. doi: 10.1097/01.psy.0000149259.72488.09. PMID 15784782
- [Derived] Lee SM, Te S, Breen EC, Olmstead R, Irwin MR, Cho JH. Circulating versus lipopolysaccharide-induced inflammatory markers as correlates of subthreshold depressive symptoms in older adults. World J Biol Psychiatry. 2020 Oct;21(8):634-641. doi: 10.1080/15622975.2019.1671608. Epub 2019 Oct 9. PMID 31552779
- [Derived] Carroll JE, Seeman TE, Olmstead R, Melendez G, Sadakane R, Bootzin R, Nicassio P, Irwin MR. Improved sleep quality in older adults with insomnia reduces biomarkers of disease risk: pilot results from a randomized controlled comparative efficacy trial. Psychoneuroendocrinology. 2015 May;55:184-92. doi: 10.1016/j.psyneuen.2015.02.010. Epub 2015 Feb 25. PMID 25770704
- [Derived] Irwin MR, Olmstead R, Breen EC, Witarama T, Carrillo C, Sadeghi N, Arevalo JM, Ma J, Nicassio P, Bootzin R, Cole S. Cognitive behavioral therapy and tai chi reverse cellular and genomic markers of inflammation in late-life insomnia: a randomized controlled trial. Biol Psychiatry. 2015 Nov 15;78(10):721-9. doi: 10.1016/j.biopsych.2015.01.010. Epub 2015 Feb 4. PMID 25748580
- [Derived] Irwin MR, Olmstead R, Carrillo C, Sadeghi N, Breen EC, Witarama T, Yokomizo M, Lavretsky H, Carroll JE, Motivala SJ, Bootzin R, Nicassio P. Cognitive behavioral therapy vs. Tai Chi for late life insomnia and inflammatory risk: a randomized controlled comparative efficacy trial. Sleep. 2014 Sep 1;37(9):1543-52. doi: 10.5665/sleep.4008. PMID 25142571